CLINICAL TRIAL: NCT04334148
Title: Healthcare Worker Exposure Response and Outcomes of Hydroxychloroquine Trial (HERO-HCQ Trial)
Brief Title: Healthcare Worker Exposure Response and Outcomes of Hydroxychloroquine
Acronym: HERO-HCQ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Hernandez (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00105274
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: Hydroxychloroquine; Coronavirus Infections; Novel Coronavirus; Protective agents; Prophylaxis; Chemoprophylaxis; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome, Adult; Acute Lung Injury; Virus Diseases; Lung Diseases; Respiratory Tract Diseases; Respiration Disorders; Lung Injury; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Respiratory Tract Infections; Antimalarials; Antiprotozoal Agents; Antiparasitic Agents; Anti-Infective Agents; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Antirheumatic Agents; Chloroquine; Chloroquine diphosphate
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Respiratory Distress Syndrome; Acute Lung Injury; Virus Diseases; Lung Diseases; Respiratory Tract Diseases; Respiration Disorders; Lung Injury; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Respiratory Tract Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine tablet 600mg bid loading dose on day 1 followed by 400mg on days 2-30.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — oral self administered tablet
  Other Names: Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo oral tablet — oral self administered tablet
  Arms: Placebo

SUMMARY:
This is a double blind, placebo controlled study in approximately 2,000 health care workers at risk for being exposed to COVID-19. Eligible participants will be randomly assigned (1:1) to either treatment group (HCQ) or placebo in a double-blind fashion. Course of treatment is 30 days.

DETAILED DESCRIPTION:
This is a double blind, placebo controlled study in approximately 2,000 health care workers at risk for being exposed to COVID-19. Eligible participants will be randomly assigned (1:1) to either treatment group (HCQ) or placebo in a double-blind fashion. After enrollment, baseline assessments will include nasopharyngeal swab for COVID-19 and a blood sample to detect seroconversion to COVID-19. For convenience, follow-up will be performed weekly through a direct to participant portal. A call center will provide support for any missed visits. Follow-up includes screening for any COVID-19 clinical infections, other respiratory infections, clinical events, adverse events, and Quality of Life (QoL) assessments. Course of treatment is 30 days. Participants are followed via survey weekly. At the end of treatment participants will return for repeat nasopharyngeal swab for COVID-19 and a blood sample to detect seroconversion to COVID-19. There will be one last contact at 8 weeks (2 months) from baseline.

ELIGIBILITY:
Inclusion:

* Completed Informed Consent
* Age ≥ 18 years old
* Currently working in any environment in which there is a risk of exposure to patients with COVID-19 infections ("healthcare worker")

Exclusion Criteria:

* Prior diagnosis of COVID-19 infection
* Participation in another COVID-19 prophylaxis trial within 30 days of consent
* Respiratory illness with new-onset fever (Temperature > 100°F) or ongoing cough or dyspnea within 14 days
* Known allergy to HCQ or chloroquine
* Congenital prolonged QT syndrome
* Current or planned use of QT prolonging drugs (e.g. procainamide, disopyramide, mexiletine, flecainide, propafenone, amiodarone, sotalol, cimetidine, dronedarone, dofetilide, levofloxacin, ciprofloxacin, moxifloxacin) and other contraindicated medications
* End stage renal disease
* Pre-existing retinopathy
* Current or planned use of Hydroxychloroquine (study drug) for any indication

Current or planned use of the following for treatment or prevention of COVID-19 infection:

* Chloroquine
* Azithromycin

  * Known cirrhosis or severe liver disease
  * History of severe skin reactions such as Steven-Johnson syndrome, toxic epidermal necrolysis
  * History of psoriasis or porphyria
  * Ventricular arrhythmias requiring medical treatment
  * Severe coronary artery disease or heart failure/cardiomyopathy with ongoing symptoms
  * Current or planned use of use of anti-seizure drugs
  * History of Glucose-6-phosphate dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1360 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, Principal Investigator — Duke University
Locations (34):
- United States (34):
  - Children's Hospital Colorado/University of Colorado Denver, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - University of Florida Health Central Florida, Leesburg, Florida
  - University of Miami Florida, Miami, Florida
  - Advent Health, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern Medicine, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Allina Health, Minneapolis, Minnesota
  - Mayo Clinic Hospital Rochester, Rochester, Minnesota
  - University of Missouri-Columbia, Columbia, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Columbia University, Irving Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor Scott & White Medical Center-Temple, Temple, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Marshfield Clinic Health System, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Plan description: HERO-HCQ is funded by PCORI, the Patient-Centered Outcomes Research Institute. PCORI calls for the researchers PCORI funds to share their data sets and documentation for reanalysis and reuse. The policy advances PCORI's commitment to open science by encouraging use of data from the studies it funds to allow other researchers to verify and build on those findings to generate new evidence available to healthcare decision makers.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: July 2022
Access Criteria: Individual investigators or teams of investigators seeking access to data from PCORI-funded studies must complete and submit a data request form to a PCORI-designated repository. The repository will independently review requests for data based on qualifications of the data requestors and the scientific merit of the request (see below). If the data request is approved, the data requestor's institution must enter into a Data Use Agreement (DUA) with the repository. More information is available here https://www.pcori.org/about-us/governance/policy-data-management-and-data-sharing
URL: http://www.pcori.org

REFERENCES:
- [Derived] Naggie S, Milstone A, Castro M, Collins SP, Lakshmi S, Anderson DJ, Cahuayme-Zuniga L, Turner KB, Cohen LW, Currier J, Fraulo E, Friedland A, Garg J, George A, Mulder H, Olson RE, O'Brien EC, Rothman RL, Shenkman E, Shostak J, Woods CW, Anstrom KJ, Hernandez AF; HERO Research Program. Hydroxychloroquine for pre-exposure prophylaxis of COVID-19 in health care workers: a randomized, multicenter, placebo-controlled trial Healthcare Worker Exposure Response and Outcomes of Hydroxychloroquine (HERO-HCQ). Int J Infect Dis. 2023 Apr;129:40-48. doi: 10.1016/j.ijid.2023.01.019. Epub 2023 Jan 20. PMID 36682681

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant was excluded from analysis population if they had a positive nasal swab test at baseline visit. This occurred to 1 participant assigned to the placebo group.
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 683 | 677
Completed | 683 | 676
Not Completed | 0 | 1
Not completed — positive nasal swab at baseline | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 683 | 676 | 1359
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.9) | 43.1 (11.2) | 43.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 442 | 446 | 888
  Male | 241 | 230 | 471
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 40 | 79
  Not Hispanic or Latino | 639 | 629 | 1268
  Unknown or Not Reported | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 28 | 27 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 18 | 23 | 41
  White | 624 | 610 | 1234
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 683 | 676 | 1359

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Infection With COVID-19 Infection
Description: This measure was a combination of confirmed infection and suspected infection. Confirmed clinical infection was defined as new-onset of fever or cough or dyspnea AND confirmed COVID-19 positive test result via local PCRI testing. Suspected infection was defined as new-onset fever or cough or dyspnea without local PCR testing due to local restrictions and/or testing policies.
Time Frame: 30 days
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 683 | 676
Participants | 41 | 53
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Other; p = 0.200, Fisher Exact

2. Secondary Outcome: Number of Participants With COVID-19 Viral Shedding
Description: Number of participants with COVID-19 infection shedding via Covance swab PCR testing
Time Frame: 30 days
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 683 | 676
Participants | 2 | 2
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Other; p = 1.0, Regression, Linear

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) or Hydroxychloroquine-Associated Events of Special Interest (EOSIs)
Description: Safety and Tolerability as determined by subject reported serious adverse events (SAEs) and hydroxychloroquine-associated events of special interest. EOSIs include: arrhythmias (ventricular), hepatic failure, bone marrow failure, aplastic anemia, prolonged QT interval, angioedema, dermatitis exfoliative, acute generalized exanthematous pustulosis, psychosis, suicidal ideation, seizure, methemoglobinemia.
Time Frame: 30 days
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 683 | 676
Participants | 7 | 8
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority; p = 0.802, Chi-squared

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Hydroxychloroquine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/683 | 0/677
Serious Adverse Events (participants affected / at risk) | 3/683 | 2/677
Other Adverse Events (participants affected / at risk) | 0/683 | 0/677
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=683) | Placebo (N=677)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol Use Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was underpowered to detect a small treatment effect. The trial was novel and improved feasibility, particularly during a pandemic. Testing was not performed at all institutions per local policies in HCW. These events were defined as suspected cases and were combined with the confirmed cases in the primary outcome. This resulted in few confirmed COVID-19 infections; thus, our primary outcome was primarily suspected COVID-19 clinical infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT04334148/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT04334148/SAP_001.pdf